CLINICAL TRIAL: NCT00039871
Title: PEG-Intron Plus REBETOL for the Treatment of Subjects With Chronic Hepatitis C Who Failed to Respond to Previous Combination Therapy (Any Alpha Interferon Treatment in Combination With Ribavirin)
Brief Title: PEG-Intron Plus Rebetol Treatment of Chronic Hepatitis C Subjects Who Failed Response to Alpha-Interferon Plus Ribavirin (Study P02370)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P02370
Record Dates: First submitted 2002-06-13; First posted 2002-06-14 (Estimated); Results first posted 2008-12-11 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis; Hepatitis C, Chronic; Fibrosis; Liver Cirrhosis
MeSH Terms: conditions — Hepatitis; Hepatitis C, Chronic; Fibrosis; Liver Cirrhosis | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Overall study population (Experimental)
  Interventions: Biological: PegIntron (peginterferon alfa-2b; SCH 54031); Drug: REBETOL (ribavirin; SCH 18908)

INTERVENTIONS:
Biological: PegIntron (peginterferon alfa-2b; SCH 54031) — PegIntron (peginterferon alfa-2b) administered at a dose of 1.5 mcg/kg subcutaneously (SC) once a week (QW) for up to 48 weeks
  Other Names: SCH 54031
Drug: REBETOL (ribavirin; SCH 18908) — REBETOL (ribavirin) administered on a weight basis: 800-1400 mg/day orally (PO) for up to 48 weeks

SUMMARY:
The objective of this study is to determine the effectiveness of PEG-Intron 1.5 ug/kg/wk plus REBETOL (ribavirin) 800-1400 mg/day in adults with chronic hepatitis C with moderate to severe liver fibrosis or cirrhosis who failed to respond to previous treatment with an alpha interferon in combination with ribavirin. Patients who do not respond to PEG-Intron plus REBETOL (ribavirin) will be enrolled in a long-term maintenance study to evaluate the effectiveness of PEG-Intron monotherapy versus no treatment for the prevention of disease progression (Protocols P02569 and P02570).

ELIGIBILITY:
Inclusion Criteria:

* Age at entry 18-65
* Positive for Hepatitis C
* Nonresponder to previous treatment (minimum of 3 months) with an alpha Interferon plus ribavirin
* Liver biopsy demonstrating moderate to severe fibrosis or cirrhosis

Exclusion Criteria:

* Any cause for the liver disease other than chronic hepatitis C
* History or presence of complications of cirrhosis
* Alcohol or illicit drug use or methadone treatment within the past 2 years
* Treatment for chronic hepatitis C within the previous 6 months
* Diseases or conditions that could interfere with the subject's participation in and completion of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2333 (Actual)
Dates: Start 2002-05; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Poynard T, Munteanu M, Colombo M, Bruix J, Schiff E, Terg R, Flamm S, Moreno-Otero R, Carrilho F, Schmidt W, Berg T, McGarrity T, Heathcote EJ, Goncales F, Diago M, Craxi A, Silva M, Boparai N, Griffel L, Burroughs M, Brass C, Albrecht J. FibroTest is an independent predictor of virologic response in chronic hepatitis C patients retreated with pegylated interferon alfa-2b and ribavirin in the EPIC(3) program. J Hepatol. 2011 Feb;54(2):227-35. doi: 10.1016/j.jhep.2010.06.038. Epub 2010 Sep 15. PMID 21056496

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolled 2333; 21 subjects excluded due to Good Clinical Practice (GCP) non-compliance.
Period: Overall Study
Arm/Group | PegIntron Plus Rebetol
Started | 2312 (Enrolled 2333; 21 subjects excluded due to GCP non-compliance)
Completed | 928
Not Completed | 1384
Not completed — Adverse Event | 165
Not completed — Lost to Follow-up | 18
Not completed — Protocol Violation | 24
Not completed — Withdrawal by Subject | 97
Not completed — Did not meet eligibility criteria | 11
Not completed — Administrative | 1
Not completed — Discontinued at Week 12 per protocol | 1061
Not completed — Never entered follow-up | 7

BASELINE CHARACTERISTICS:
Arm/Group | PegIntron Plus Rebetol
Number analyzed (Participants) | 2312
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2267
  >=65 years | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 662
  Male | 1650
Hepatitis C Virus (HCV) Genotype [Number; unit: number of participants]
  Genotype 1 | 1859
  Genotype 2 | 75
  Genotype 3 | 293
  Genotype 4 | 68
  Nontypable | 8
  Missing | 9
METAVIR Fibrosis score [Number; unit: number of participants] — The METAVIR scoring system for hepatic fibrosis is as follows:
  * F0= no fibrosis
  * F1 = portal fibrosis without septa
  * F2 = portal fibrosis with few septa
  * F3= septal fibrosis without cirrhosis
  * F4= cirrhosis
  number of participants
    F1 | 2
    F2 | 658
    F3 | 676
    F4 | 974
    Missing | 2

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virologic Response (SVR) Rate
Description: Number of participants with undetectable hepatitis C virus RNA (HCV-RNA)
Time Frame: Assessed at end of 24 weeks posttreatment follow-up
Population: Participants who received at least one dose of study medication
Measure: Number; unit: Participants
Arm/Group | PegIntron Plus Rebetol
Number analyzed (Participants) | 2293
Participants | 497
Statistical Analysis 1: Comparison: PegIntron Plus Rebetol; Test type: Superiority or Other; Binomial Approximation = 0.217, 99% CI [0.195 to 0.239]

2. Secondary Outcome: Sustained Virologic Response (SVR) for Participants With Undetectable HCV-RNA at Treatment Week 12
Description: Number of participants with undetectable HCV-RNA at Treatment Week 12 who had subsequent undetectable HCV-RNA after 24 weeks of posttreatment follow-up
Time Frame: 24 weeks posttreatment
Population: Participants who had undetectable HCV-RNA at Treatment Week 12
Measure: Number; unit: Participants
Arm/Group | PegIntron Plus Rebetol
Number analyzed (Participants) | 823
Participants | 463
Statistical Analysis 1: Comparison: PegIntron Plus Rebetol; Test type: Superiority or Other; Binomial Approximation = 0.563, 95% CI [0.529 to 0.596]

3. Secondary Outcome: Sustained Virologic Response (SVR) for Participants With Detectable But ≥2 Log Drop in HCV-RNA at Treatment Week 12
Description: Number of participants with detectable HCV-RNA but ≥2 log drop from baseline in HCV-RNA at Treatment Week 12 who had subsequent undetectable HCV-RNA after 24 weeks of posttreatment follow-up
Time Frame: 24 weeks posttreatment
Population: Participants with detectable but >=2 log drop in HCV-RNA at Treatment Week 12
Measure: Number; unit: Participants
Arm/Group | PegIntron Plus Rebetol
Number analyzed (Participants) | 188
Participants | 23
Statistical Analysis 1: Comparison: PegIntron Plus Rebetol; Test type: Superiority or Other; Binomial Approximation = 0.122, 95% CI [0.076 to 0.169]

ADVERSE EVENTS:
Arm/Group | PegIntron Plus Rebetol
Serious Adverse Events (participants affected / at risk) | 200/2312
Other Adverse Events (participants affected / at risk) | 2201/2312
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PegIntron Plus Rebetol (N=2312)
ANAEMIA (Blood and lymphatic system disorders) | 4 (4)
AUTOIMMUNE THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1)
LEUKOPENIA (Blood and lymphatic system disorders) | 3 (3)
LYMPHADENOPATHY MEDIASTINAL (Blood and lymphatic system disorders) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 7 (9)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (2)
THROMBOTIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
ANGINA UNSTABLE (Cardiac disorders) | 2 (2)
ATRIAL FIBRILLATION (Cardiac disorders) | 4 (4)
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 1 (1)
CARDIAC DISORDER (Cardiac disorders) | 1 (1)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 2 (2)
MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (2)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1)
POSTINFARCTION ANGINA (Cardiac disorders) | 1 (1)
HYDROCELE (Congenital, familial and genetic disorders) | 1 (1)
DEAFNESS (Ear and labyrinth disorders) | 1 (1)
HYPOACUSIS (Ear and labyrinth disorders) | 2 (2)
MENIERE'S DISEASE (Ear and labyrinth disorders) | 1 (1)
ADRENAL MASS (Endocrine disorders) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1)
CATARACT (Eye disorders) | 2 (4)
EYE INFLAMMATION (Eye disorders) | 1 (1)
GLAUCOMA (Eye disorders) | 1 (1)
RETINAL ARTERY STENOSIS (Eye disorders) | 1 (2)
RETINAL HAEMORRHAGE (Eye disorders) | 1 (1)
VISION BLURRED (Eye disorders) | 2 (3)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (3)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (2)
ANAL FISSURE (Gastrointestinal disorders) | 1 (1)
APPENDICITIS PERFORATED (Gastrointestinal disorders) | 1 (2)
ASCITES (Gastrointestinal disorders) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 3 (3)
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1)
EROSIVE DUODENITIS (Gastrointestinal disorders) | 1 (1)
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 1 (1)
HAEMATEMESIS (Gastrointestinal disorders) | 1 (1)
HAEMORRHOIDS (Gastrointestinal disorders) | 2 (2)
INGUINAL HERNIA (Gastrointestinal disorders) | 2 (2)
MALLORY-WEISS SYNDROME (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 4 (4)
OESOPHAGEAL ULCER (Gastrointestinal disorders) | 1 (1)
OESOPHAGITIS (Gastrointestinal disorders) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 2 (2)
SALIVARY GLAND CALCULUS (Gastrointestinal disorders) | 1 (1)
UMBILICAL HERNIA (Gastrointestinal disorders) | 1 (1)
VARICES OESOPHAGEAL (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 3 (3)
VOMITING PROJECTILE (Gastrointestinal disorders) | 1 (1)
ASTHENIA (General disorders) | 3 (3)
CHEST PAIN (General disorders) | 8 (8)
DISEASE PROGRESSION (General disorders) | 2 (2)
FATIGUE (General disorders) | 2 (2)
MULTI-ORGAN FAILURE (General disorders) | 2 (2)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1)
PYREXIA (General disorders) | 4 (4)
CHOLECYSTITIS (Hepatobiliary disorders) | 2 (2)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 4 (4)
CHOLELITHIASIS (Hepatobiliary disorders) | 4 (4)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 (1)
HEPATIC FAILURE (Hepatobiliary disorders) | 1 (1)
HEPATIC LESION (Hepatobiliary disorders) | 1 (1)
HEPATORENAL SYNDROME (Hepatobiliary disorders) | 1 (1)
HYDROCHOLECYSTIS (Hepatobiliary disorders) | 1 (1)
JAUNDICE (Hepatobiliary disorders) | 1 (1)
APPENDICITIS (Infections and infestations) | 6 (6)
BACTERAEMIA (Infections and infestations) | 1 (1)
BOUTONNEUSE FEVER (Infections and infestations) | 2 (2)
BRONCHITIS (Infections and infestations) | 1 (1)
BRONCHOPNEUMONIA (Infections and infestations) | 1 (1)
CELLULITIS (Infections and infestations) | 7 (7)
CELLULITIS STAPHYLOCOCCAL (Infections and infestations) | 1 (1)
CERVICITIS (Infections and infestations) | 1 (1)
DIVERTICULITIS (Infections and infestations) | 2 (3)
ERYSIPELAS (Infections and infestations) | 1 (1)
ESCHERICHIA SEPSIS (Infections and infestations) | 1 (1)
FURUNCLE (Infections and infestations) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 4 (4)
GASTROENTERITIS SALMONELLA (Infections and infestations) | 2 (2)
LEPROSY (Infections and infestations) | 1 (1)
LOBAR PNEUMONIA (Infections and infestations) | 2 (2)
LUNG ABSCESS (Infections and infestations) | 1 (1)
LUNG INFECTION (Infections and infestations) | 1 (1)
NECROTISING FASCIITIS (Infections and infestations) | 1 (1)
OTITIS MEDIA (Infections and infestations) | 1 (1)
PELVIC INFLAMMATORY DISEASE (Infections and infestations) | 1 (1)
PERITONEAL ABSCESS (Infections and infestations) | 1 (1)
PERITONITIS BACTERIAL (Infections and infestations) | 2 (3)
PNEUMONIA (Infections and infestations) | 10 (10)
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 2 (2)
PYELONEPHRITIS ACUTE (Infections and infestations) | 2 (2)
RENAL ABSCESS (Infections and infestations) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1)
SEPSIS SYNDROME (Infections and infestations) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 1 (1)
SINUSITIS (Infections and infestations) | 1 (1)
STAPHYLOCOCCAL ABSCESS (Infections and infestations) | 1 (1)
SUPERINFECTION (Infections and infestations) | 1 (1)
TRACHEOBRONCHITIS (Infections and infestations) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1)
ACCIDENT AT WORK (Injury, poisoning and procedural complications) | 1 (1)
ANIMAL BITE (Injury, poisoning and procedural complications) | 1 (1)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
ARTHROPOD STING (Injury, poisoning and procedural complications) | 1 (1)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
CONCUSSION (Injury, poisoning and procedural complications) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1)
EXTRADURAL HAEMATOMA (Injury, poisoning and procedural complications) | 2 (2)
EYE INJURY (Injury, poisoning and procedural complications) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 3 (3)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
FOREIGN BODY TRAUMA (Injury, poisoning and procedural complications) | 1 (1)
HAND FRACTURE (Injury, poisoning and procedural complications) | 2 (2)
HEAD INJURY (Injury, poisoning and procedural complications) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
INJURY (Injury, poisoning and procedural complications) | 1 (1)
INTENTIONAL OVERDOSE (Injury, poisoning and procedural complications) | 1 (1)
JAW FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 2 (2)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 2 (2)
OVERDOSE (Injury, poisoning and procedural complications) | 2 (3)
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 1 (1)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 6 (6)
SKIN LACERATION (Injury, poisoning and procedural complications) | 1 (1)
SKULL FRACTURED BASE (Injury, poisoning and procedural complications) | 2 (3)
STENT OCCLUSION (Injury, poisoning and procedural complications) | 1 (1)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 (1)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 (1)
BLOOD PRESSURE ORTHOSTATIC (Investigations) | 1 (1)
HAEMOGLOBIN DECREASED (Investigations) | 3 (4)
ANOREXIA (Metabolism and nutrition disorders) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 3 (3)
DIABETES MELLITUS INSULIN-DEPENDENT (Metabolism and nutrition disorders) | 1 (2)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1 (1)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 2 (2)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 1 (1)
BILIARY ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
HEPATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
RENAL CELL CARCINOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CEREBELLAR INFARCTION (Nervous system disorders) | 1 (1)
CEREBRAL INFARCTION (Nervous system disorders) | 2 (2)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2 (2)
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 1 (1)
COMA (Nervous system disorders) | 3 (3)
CONVULSION (Nervous system disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (2)
ENCEPHALOPATHY (Nervous system disorders) | 1 (1)
FACIAL PALSY (Nervous system disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 2 (2)
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 1 (1)
HYDROCEPHALUS (Nervous system disorders) | 1 (1)
HYPOAESTHESIA (Nervous system disorders) | 1 (1)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 3 (3)
MIGRAINE (Nervous system disorders) | 1 (1)
PARAESTHESIA (Nervous system disorders) | 1 (1)
QUADRIPARESIS (Nervous system disorders) | 1 (1)
RADICULOPATHY (Nervous system disorders) | 1 (1)
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 (1)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 2 (2)
SYNCOPE (Nervous system disorders) | 4 (4)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 2 (3)
VISUAL FIELD DEFECT (Nervous system disorders) | 2 (3)
FOETAL GROWTH RETARDATION (Pregnancy, puerperium and perinatal conditions) | 1 (1)
INTRA-UTERINE DEATH (Pregnancy, puerperium and perinatal conditions) | 1 (1)
RETROPLACENTAL HAEMATOMA (Pregnancy, puerperium and perinatal conditions) | 1 (1)
ACUTE PSYCHOSIS (Psychiatric disorders) | 1 (1)
AGGRESSION (Psychiatric disorders) | 1 (1)
BIPOLAR DISORDER (Psychiatric disorders) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1)
DEPENDENCE (Psychiatric disorders) | 1 (1)
DEPRESSION (Psychiatric disorders) | 10 (10)
HALLUCINATION (Psychiatric disorders) | 3 (3)
HALLUCINATION, AUDITORY (Psychiatric disorders) | 1 (1)
HALLUCINATION, VISUAL (Psychiatric disorders) | 1 (1)
HOMICIDAL IDEATION (Psychiatric disorders) | 1 (1)
MOOD SWINGS (Psychiatric disorders) | 1 (1)
PERSECUTORY DELUSION (Psychiatric disorders) | 1 (1)
PHOBIA (Psychiatric disorders) | 1 (1)
PSYCHOTIC DISORDER (Psychiatric disorders) | 3 (3)
SUICIDAL IDEATION (Psychiatric disorders) | 8 (8)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1)
CALCULUS URETERIC (Renal and urinary disorders) | 1 (1)
CALCULUS URINARY (Renal and urinary disorders) | 1 (1)
DYSURIA (Renal and urinary disorders) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 2 (2)
RENAL COLIC (Renal and urinary disorders) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 2 (2)
RENAL MASS (Renal and urinary disorders) | 1 (1)
ADENOMYOSIS (Reproductive system and breast disorders) | 1 (1)
MENORRHAGIA (Reproductive system and breast disorders) | 1 (1)
TESTICULAR NECROSIS (Reproductive system and breast disorders) | 1 (1)
VARICOCELE (Reproductive system and breast disorders) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 (3)
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1 (1)
ECZEMA ASTEATOTIC (Skin and subcutaneous tissue disorders) | 1 (1)
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 1 (1)
SKIN LESION (Skin and subcutaneous tissue disorders) | 1 (1)
MISCARRIAGE OF PARTNER (Social circumstances) | 1 (1)
PREGNANCY OF PARTNER (Social circumstances) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2)
HAEMATOMA (Vascular disorders) | 3 (3)
HAEMORRHAGE (Vascular disorders) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1)
THROMBOSIS (Vascular disorders) | 1 (1)
VARICOSE VEIN (Vascular disorders) | 1 (1)
VASCULAR PSEUDOANEURYSM (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PegIntron Plus Rebetol (N=2312)
ANAEMIA (Blood and lymphatic system disorders) | 372 (721)
LEUKOPENIA (Blood and lymphatic system disorders) | 239 (538)
NEUTROPENIA (Blood and lymphatic system disorders) | 455 (1271)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 174 (436)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 155 (206)
DIARRHOEA (Gastrointestinal disorders) | 342 (486)
DRY MOUTH (Gastrointestinal disorders) | 145 (155)
DYSPEPSIA (Gastrointestinal disorders) | 129 (150)
NAUSEA (Gastrointestinal disorders) | 587 (925)
VOMITING (Gastrointestinal disorders) | 210 (281)
ASTHENIA (General disorders) | 496 (1086)
CHILLS (General disorders) | 510 (768)
FATIGUE (General disorders) | 759 (1108)
INFLUENZA LIKE ILLNESS (General disorders) | 493 (1285)
INJECTION SITE ERYTHEMA (General disorders) | 237 (326)
INJECTION SITE REACTION (General disorders) | 120 (128)
IRRITABILITY (General disorders) | 398 (566)
PYREXIA (General disorders) | 900 (2406)
WEIGHT DECREASED (Investigations) | 154 (191)
ANOREXIA (Metabolism and nutrition disorders) | 286 (365)
DECREASED APPETITE (Metabolism and nutrition disorders) | 202 (222)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 391 (686)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 172 (216)
MYALGIA (Musculoskeletal and connective tissue disorders) | 714 (2249)
DIZZINESS (Nervous system disorders) | 251 (358)
HEADACHE (Nervous system disorders) | 938 (2801)
ANXIETY (Psychiatric disorders) | 212 (289)
DEPRESSION (Psychiatric disorders) | 281 (383)
INSOMNIA (Psychiatric disorders) | 519 (772)
COUGH (Respiratory, thoracic and mediastinal disorders) | 374 (447)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 250 (313)
ALOPECIA (Skin and subcutaneous tissue disorders) | 392 (417)
DRY SKIN (Skin and subcutaneous tissue disorders) | 196 (220)
PRURITUS (Skin and subcutaneous tissue disorders) | 358 (471)
RASH (Skin and subcutaneous tissue disorders) | 224 (297)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less